CLINICAL TRIAL: NCT00269087
Title: Clinical Evaluation of GW815SF for Chronic Obstructive Pulmonary Disease (Chronic Bronchitis, Emphysema)" A Long-term Treatment Study of GW815SF50/500µg in Chronic Obstructive Pulmonary Disease -
Brief Title: GW815SF For Chronic Obstructive Pulmonary Disease (Chronic Bronchitis, Emphysema)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCO100648
Record Dates: First submitted 2005-12-21; First posted 2005-12-23 (Estimated); Results first posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2018-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Bronchitis; COPD; Emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema | interventions — Fluticasone

INTERVENTIONS:
Drug: fluticasone propionate/salmeterol combination DISKUS

SUMMARY:
This study evaluates the safety of medicine on COPD (Chronic Obstructive Pulmonary Disease). This study will last up to 56 weeks, and subjects will visit the clinic 16 times. Subjects will be given breathing tests, and will record their breathing symptoms daily on diary cards.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of COPD.

Exclusion criteria:

* Diagnosis of asthma or an uncontrolled medical condition or respiratory disorder other than COPD.
* Other inclusion and exclusion criteria will be evaluated at the first study visit.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2005-01-28; Primary Completion 2006-10-01 (Actual); Study Completion 2006-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Japan (4):
  - GSK Investigational Site, Kodaira
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
- GSK Investigational Site

REFERENCES:
- [Background] This study has not been published in the scientific literature.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A study was conducted at 20 centers in Japan from 28 December 2004 to 25 October 2006.
Pre-assignment Details: The study period consisted of 2-week run-in period (could be extended up to 4 weeks). Total 174 participants entered into the study, of which 127 participants were screened and entered into run-in phase. Five participants withdrew from the study during run-in phase and total 122 participants received study medication.
Groups:
- GW815SF 50/500 µg: Participants received one inhalation of GW815SF 50/500 micrograms (µg) (50 µg salmeterol and 500 µg fluticasone propionate) twice daily for 52 weeks. Participants also received Salbutamol sulfate aerosol as a rescue medication on an as-needed basis.
Period: Overall Study
Arm/Group | GW815SF 50/500 µg
Started | 122
Completed | 88
Not Completed | 34
Not completed — Adverse Event | 20
Not completed — Withdrawal by Subject | 1
Not completed — Exacerbation of COPD | 13

BASELINE CHARACTERISTICS:
Groups:
- GW815SF 50/500 µg: Participants received one inhalation of GW815SF 50/500 µg (50 µg salmeterol and 500 µg fluticasone propionate) twice daily for 52 weeks. Participants also received Salbutamol sulfate aerosol as a rescue medication on an as-needed basis.
Arm/Group | GW815SF 50/500 µg
Number analyzed (Participants) | 122
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.2 (6.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 116
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 122
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Events (AEs) and Serious AEs (SAEs)
Description: AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE include adverse events that result in any of the following outcomes: death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: Up to Week 56
Population: Safety Population included all participants who had received an investigational product even for once.
Measure: Count of Participants; unit: Participants
Arm/Group | GW815SF 50/500 µg
Number analyzed (Participants) | 122
Participants
  Any AEs | 120
  Any SAEs | 27

2. Secondary Outcome: Number of Participants With Abnormal (Outliers From the Normal Range) Hematology Parameters
Description: Hematology parameters: Red blood cells (RBC), Hemoglobin (Hb), Hematocrit, Platelet count (PC), White blood cells (WBC), Basophils, Eosinophils, Neutrophils, Lymphocytes and Monocytes were presented as the outliers from the normal range as > upper limit and < lower limit. Only number of participants with hematology values outside normal range were presented.
Time Frame: Up to Week 56
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GW815SF 50/500 µg
Number analyzed (Participants) | 122
Participants
  RBC, Baseline, < lower limit | 30
  RBC, Week 4, < lower limit: number analyzed (Participants) | 121
  RBC, Week 4, < lower limit | 36
  RBC, Week 12, < lower limit: number analyzed (Participants) | 113
  RBC, Week 12, < lower limit | 36
  RBC, Week 24, > upper limit: number analyzed (Participants) | 106
  RBC, Week 24, > upper limit | 1
  RBC, Week 24, < lower limit: number analyzed (Participants) | 106
  RBC, Week 24, < lower limit | 21
  RBC, Week 36, > upper limit: number analyzed (Participants) | 95
  RBC, Week 36, > upper limit | 1
  RBC, Week 36, < lower limit: number analyzed (Participants) | 95
  RBC, Week 36, < lower limit | 22
  RBC, Week 52/Withdrawal, > upper limit: number analyzed (Participants) | 113
  RBC, Week 52/Withdrawal, > upper limit | 1
  RBC, Week 52/Withdrawal, < lower limit: number analyzed (Participants) | 113
  RBC, Week 52/Withdrawal, < lower limit | 33
  Hb, Baseline, > upper limit | 1
  Hb, Baseline, < lower limit | 15
  Hb, Week 4, < lower limit: number analyzed (Participants) | 121
  Hb, Week 4, < lower limit | 20
  Hb, Week 12, < lower limit: number analyzed (Participants) | 113
  Hb, Week 12, < lower limit | 20
  Hb, Week 24, < lower limit: number analyzed (Participants) | 106
  Hb, Week 24, < lower limit | 13
  Hb, Week 36, < lower limit: number analyzed (Participants) | 95
  Hb, Week 36, < lower limit | 14
  Hb, Week 52/Withdrawal, <lower limit: number analyzed (Participants) | 113
  Hb, Week 52/Withdrawal, <lower limit | 27
  Hematocrit, Baseline, > upper limit | 4
  Hematocrit, Baseline, < lower limit | 10
  Hematocrit, Week 4, > upper limit: number analyzed (Participants) | 121
  Hematocrit, Week 4, > upper limit | 1
  Hematocrit, Week 4, < lower limit: number analyzed (Participants) | 121
  Hematocrit, Week 4, < lower limit | 13
  Hematocrit, Week 12, > upper limit: number analyzed (Participants) | 113
  Hematocrit, Week 12, > upper limit | 1
  Hematocrit, Week 12, < lower limit: number analyzed (Participants) | 113
  Hematocrit, Week 12, < lower limit | 13
  Hematocrit, Week 24, > upper limit: number analyzed (Participants) | 106
  Hematocrit, Week 24, > upper limit | 1
  Hematocrit, Week 24, < lower limit: number analyzed (Participants) | 106
  Hematocrit, Week 24, < lower limit | 9
  Hematocrit, Week 36, < lower limit: number analyzed (Participants) | 95
  Hematocrit, Week 36, < lower limit | 12
  Hematocrit,Week 52/Withdrawal,< lower limit: number analyzed (Participants) | 113
  Hematocrit,Week 52/Withdrawal,< lower limit | 17
  PC, Baseline, > upper limit | 3
  PC, Baseline, < lower limit | 8
  PC, Week 4, > upper limit: number analyzed (Participants) | 121
  PC, Week 4, > upper limit | 1
  PC, Week 4, < lower limit: number analyzed (Participants) | 121
  PC, Week 4, < lower limit | 7
  PC, Week 12, > upper limit: number analyzed (Participants) | 113
  PC, Week 12, > upper limit | 7
  PC, Week 12, < lower limit: number analyzed (Participants) | 113
  PC, Week 12, < lower limit | 6
  PC, Week 24, > upper limit: number analyzed (Participants) | 105
  PC, Week 24, > upper limit | 5
  PC, Week 24, < lower limit: number analyzed (Participants) | 105
  PC, Week 24, < lower limit | 4
  PC, Week 36, > upper limit: number analyzed (Participants) | 95
  PC, Week 36, > upper limit | 2
  PC, Week 36, < lower limit: number analyzed (Participants) | 95
  PC, Week 36, < lower limit | 6
  PC, Week 52/Withdrawal, > upper limit: number analyzed (Participants) | 112
  PC, Week 52/Withdrawal, > upper limit | 4
  PC, Week 52/Withdrawal, < lower limit: number analyzed (Participants) | 112
  PC, Week 52/Withdrawal, < lower limit | 2
  WBC, Baseline, > upper limit | 4
  WBC, Baseline, < lower limit | 2
  WBC, Week 4, > upper limit: number analyzed (Participants) | 121
  WBC, Week 4, > upper limit | 3
  WBC, Week 4, < lower limit: number analyzed (Participants) | 121
  WBC, Week 4, < lower limit | 3
  WBC, Week 12, > upper limit: number analyzed (Participants) | 113
  WBC, Week 12, > upper limit | 2
  WBC, Week 24, > upper limit: number analyzed (Participants) | 106
  WBC, Week 24, > upper limit | 5
  WBC, Week 24, < lower limit: number analyzed (Participants) | 106
  WBC, Week 24, < lower limit | 1
  WBC, Week 36, > upper limit: number analyzed (Participants) | 95
  WBC, Week 36, > upper limit | 5
  WBC, Week 36, < lower limit: number analyzed (Participants) | 95
  WBC, Week 36, < lower limit | 2
  WBC, Week 52/Withdrawal, > upper limit: number analyzed (Participants) | 113
  WBC, Week 52/Withdrawal, > upper limit | 7
  Basophils, Baseline, > upper limit | 1
  Basophils, Week 4, > upper limit: number analyzed (Participants) | 121
  Basophils, Week 4, > upper limit | 1
  Basophils, Week 12, > upper limit: number analyzed (Participants) | 113
  Basophils, Week 12, > upper limit | 4
  Basophils, Week 36, > upper limit: number analyzed (Participants) | 95
  Basophils, Week 36, > upper limit | 1
  Basophils, Week 52/Withdrawal, > upper limit: number analyzed (Participants) | 113
  Basophils, Week 52/Withdrawal, > upper limit | 2
  Eosinophils, Baseline, > upper limit | 17
  Eosinophils, Week 4, > upper limit: number analyzed (Participants) | 121
  Eosinophils, Week 4, > upper limit | 10
  Eosinophils, Week 12, > upper limit: number analyzed (Participants) | 113
  Eosinophils, Week 12, > upper limit | 10
  Eosinophils, Week 24, > upper limit: number analyzed (Participants) | 106
  Eosinophils, Week 24, > upper limit | 8
  Eosinophils, Week 36, > upper limit: number analyzed (Participants) | 95
  Eosinophils, Week 36, > upper limit | 8
  Eosinophils,Week 52/Withdrawal,> upper limit: number analyzed (Participants) | 113
  Eosinophils,Week 52/Withdrawal,> upper limit | 10
  Neutrophils, Baseline, > upper limit | 5
  Neutrophils, Baseline, < lower limit | 5
  Neutrophils, Week 4, > upper limit: number analyzed (Participants) | 121
  Neutrophils, Week 4, > upper limit | 7
  Neutrophils, Week 4, < lower limit: number analyzed (Participants) | 121
  Neutrophils, Week 4, < lower limit | 3
  Neutrophils, Week 12, > upper limit: number analyzed (Participants) | 113
  Neutrophils, Week 12, > upper limit | 6
  Neutrophils, Week 24, > upper limit: number analyzed (Participants) | 106
  Neutrophils, Week 24, > upper limit | 15
  Neutrophils, Week 36, > upper limit: number analyzed (Participants) | 95
  Neutrophils, Week 36, > upper limit | 9
  Neutrophils, Week 36, < lower limit: number analyzed (Participants) | 95
  Neutrophils, Week 36, < lower limit | 2
  Neutrophils,Week 52/Withdrawal,>upper limit: number analyzed (Participants) | 113
  Neutrophils,Week 52/Withdrawal,>upper limit | 11
  Neutrophils,Week 52/Withdrawal,< lower limit: number analyzed (Participants) | 113
  Neutrophils,Week 52/Withdrawal,< lower limit | 1
  Lymphocytes, Baseline, > upper limit | 2
  Lymphocytes, Baseline, < lower limit | 10
  Lymphocytes, Week 4, < lower limit: number analyzed (Participants) | 121
  Lymphocytes, Week 4, < lower limit | 16
  Lymphocytes, Week 12, < lower limit: number analyzed (Participants) | 113
  Lymphocytes, Week 12, < lower limit | 17
  Lymphocytes, Week 24, < lower limit: number analyzed (Participants) | 106
  Lymphocytes, Week 24, < lower limit | 25
  Lymphocytes, Week 36, < lower limit: number analyzed (Participants) | 95
  Lymphocytes, Week 36, < lower limit | 16
  Lymphocytes,Week 52/Withdrawal,< lower limit: number analyzed (Participants) | 113
  Lymphocytes,Week 52/Withdrawal,< lower limit | 19
  Monocytes, Baseline, > upper limit | 31
  Monocytes, Week 4, > upper limit: number analyzed (Participants) | 121
  Monocytes, Week 4, > upper limit | 47
  Monocytes, Week 12, > upper limit: number analyzed (Participants) | 113
  Monocytes, Week 12, > upper limit | 37
  Monocytes, Week 24, > upper limit: number analyzed (Participants) | 106
  Monocytes, Week 24, > upper limit | 25
  Monocytes, Week 36, > upper limit: number analyzed (Participants) | 95
  Monocytes, Week 36, > upper limit | 28
  Monocytes, wEEK 52/Withdrawal,> upper limit: number analyzed (Participants) | 113
  Monocytes, wEEK 52/Withdrawal,> upper limit | 14

3. Secondary Outcome: Number of Participants With Abnormal (Outliers From the Normal Range) Clinical Chemistry Parameters
Description: Clinical chemistry parameters: Total bilirubin (TB), Alkaline phosphatase (Al-P), Alanine aminotransferase (ALT), Asparate aminotransferase (AST), Gamma-glutamyl transpeptidase (GTP), Lactate dehydrogenase (LDH), Total cholesterol (TC), Glucose, Creatinine, Blood urea nitrogen (BUN), Uric acid (UA), Sodium (Na), Potassium (K), Chloride (Cl) and Calcium (Ca) were presented as the outliers from the normal range as > upper limit and < lower limit. Only number of participants with clinical chemistry values outside normal range were presented.
Time Frame: Up to Week 56
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GW815SF 50/500 µg
Number analyzed (Participants) | 122
Participants
  TB, Baseline, > upper limit | 1
  TB, Week 4, > upper limit: number analyzed (Participants) | 121
  TB, Week 4, > upper limit | 2
  TB, Week 12, > upper limit: number analyzed (Participants) | 113
  TB, Week 12, > upper limit | 3
  TB, Week 12, < lower limit: number analyzed (Participants) | 113
  TB, Week 12, < lower limit | 1
  TB, Week 24, > upper limit: number analyzed (Participants) | 106
  TB, Week 24, > upper limit | 5
  TB, Week 36, > upper limit: number analyzed (Participants) | 95
  TB, Week 36, > upper limit | 2
  TB, Week 36, < lower limit: number analyzed (Participants) | 95
  TB, Week 36, < lower limit | 1
  TB, Week 52/ withdrawal, > upper limit: number analyzed (Participants) | 114
  TB, Week 52/ withdrawal, > upper limit | 4
  AL-P, Baseline, > upper limit | 18
  AL-P, Week 4, > upper limit: number analyzed (Participants) | 121
  AL-P, Week 4, > upper limit | 15
  AL-P, Week 12, > upper limit: number analyzed (Participants) | 113
  AL-P, Week 12, > upper limit | 15
  AL-P, Week 24, > upper limit: number analyzed (Participants) | 106
  AL-P, Week 24, > upper limit | 18
  AL-P, Week 24, < lower limit: number analyzed (Participants) | 106
  AL-P, Week 24, < lower limit | 1
  AL-P, Week 36, > upper limit: number analyzed (Participants) | 95
  AL-P, Week 36, > upper limit | 12
  AL-P, Week 52/ withdrawal, > upper limit: number analyzed (Participants) | 114
  AL-P, Week 52/ withdrawal, > upper limit | 13
  ALT, Baseline, > upper limit | 5
  ALT, Week 4, > upper limit: number analyzed (Participants) | 121
  ALT, Week 4, > upper limit | 4
  ALT, Week 12, > upper limit: number analyzed (Participants) | 113
  ALT, Week 12, > upper limit | 7
  ALT, Week 24, > upper limit: number analyzed (Participants) | 106
  ALT, Week 24, > upper limit | 6
  ALT, Week 36, > upper limit: number analyzed (Participants) | 95
  ALT, Week 36, > upper limit | 3
  ALT, Week 52/ withdrawal, > upper limit: number analyzed (Participants) | 114
  ALT, Week 52/ withdrawal, > upper limit | 4
  AST, Baseline, > upper limit | 9
  AST, Week 4, > upper limit: number analyzed (Participants) | 121
  AST, Week 4, > upper limit | 6
  AST, Week 12, > upper limit: number analyzed (Participants) | 113
  AST, Week 12, > upper limit | 6
  AST, Week 24, > upper limit: number analyzed (Participants) | 106
  AST, Week 24, > upper limit | 9
  AST, Week 36, > upper limit: number analyzed (Participants) | 95
  AST, Week 36, > upper limit | 4
  AST, Week 52/ withdrawal, > upper limit: number analyzed (Participants) | 114
  AST, Week 52/ withdrawal, > upper limit | 5
  Gamma GTP, Baseline, > upper limit | 15
  Gamma GTP, Baseline, < lower limit | 9
  Gamma GTP, Week 4, > upper limit: number analyzed (Participants) | 121
  Gamma GTP, Week 4, > upper limit | 17
  Gamma GTP, Week 4, < lower limit: number analyzed (Participants) | 121
  Gamma GTP, Week 4, < lower limit | 10
  Gamma GTP, Week 12, > upper limit: number analyzed (Participants) | 113
  Gamma GTP, Week 12, > upper limit | 14
  Gamma GTP, Week 12, < lower limit: number analyzed (Participants) | 113
  Gamma GTP, Week 12, < lower limit | 8
  Gamma GTP, Week 24, > upper limit: number analyzed (Participants) | 106
  Gamma GTP, Week 24, > upper limit | 12
  Gamma GTP, Week 24, < lower limit: number analyzed (Participants) | 106
  Gamma GTP, Week 24, < lower limit | 8
  Gamma GTP, Week 36, > upper limit: number analyzed (Participants) | 95
  Gamma GTP, Week 36, > upper limit | 12
  Gamma GTP, Week 36, < lower limit: number analyzed (Participants) | 95
  Gamma GTP, Week 36, < lower limit | 8
  Gamma GTP,Week 52/withdrawal, > upper limit: number analyzed (Participants) | 114
  Gamma GTP,Week 52/withdrawal, > upper limit | 15
  Gamma GTP,Week 52/withdrawal, < lower limit: number analyzed (Participants) | 114
  Gamma GTP,Week 52/withdrawal, < lower limit | 10
  LDH, Baseline, > upper limit | 10
  LDH, Week 4, > upper limit: number analyzed (Participants) | 121
  LDH, Week 4, > upper limit | 11
  LDH, Week 12, > upper limit: number analyzed (Participants) | 113
  LDH, Week 12, > upper limit | 8
  LDH, Week 24, > upper limit: number analyzed (Participants) | 106
  LDH, Week 24, > upper limit | 14
  LDH, Week 36, > upper limit: number analyzed (Participants) | 95
  LDH, Week 36, > upper limit | 10
  LDH, Week 36, < lower limit: number analyzed (Participants) | 95
  LDH, Week 36, < lower limit | 1
  LDH, Week 52/ withdrawal, > upper limit: number analyzed (Participants) | 114
  LDH, Week 52/ withdrawal, > upper limit | 9
  TC, Baseline, > upper limit | 17
  TC, Baseline, < lower limit | 13
  TC, Week 4, > upper limit: number analyzed (Participants) | 121
  TC, Week 4, > upper limit | 19
  TC, Week 4, < lower limit: number analyzed (Participants) | 121
  TC, Week 4, < lower limit | 16
  TC, Week 12, > upper limit: number analyzed (Participants) | 113
  TC, Week 12, > upper limit | 21
  TC, Week 12, < lower limit: number analyzed (Participants) | 113
  TC, Week 12, < lower limit | 8
  TC, Week 24, > upper limit: number analyzed (Participants) | 106
  TC, Week 24, > upper limit | 20
  TC, Week 24, < lower limit: number analyzed (Participants) | 106
  TC, Week 24, < lower limit | 10
  TC, Week 36, > upper limit: number analyzed (Participants) | 95
  TC, Week 36, > upper limit | 22
  TC, Week 36, < lower limit: number analyzed (Participants) | 95
  TC, Week 36, < lower limit | 10
  TC, Week 52/ withdrawal, > upper limit: number analyzed (Participants) | 114
  TC, Week 52/ withdrawal, > upper limit | 27
  TC, Week 52/ withdrawal, < lower limit: number analyzed (Participants) | 114
  TC, Week 52/ withdrawal, < lower limit | 10
  Glucose, Baseline, > upper limit | 40
  Glucose, Baseline, < lower limit | 2
  Glucose, Week 4, > upper limit: number analyzed (Participants) | 121
  Glucose, Week 4, > upper limit | 42
  Glucose, Week 4, < lower limit: number analyzed (Participants) | 121
  Glucose, Week 4, < lower limit | 4
  Glucose, Week 12, > upper limit: number analyzed (Participants) | 113
  Glucose, Week 12, > upper limit | 42
  Glucose, Week 12, < lower limit: number analyzed (Participants) | 113
  Glucose, Week 12, < lower limit | 4
  Glucose, Week 24, > upper limit: number analyzed (Participants) | 106
  Glucose, Week 24, > upper limit | 31
  Glucose, Week 24, < lower limit: number analyzed (Participants) | 106
  Glucose, Week 24, < lower limit | 3
  Glucose, Week 36, > upper limit: number analyzed (Participants) | 95
  Glucose, Week 36, > upper limit | 34
  Glucose, Week 36, < lower limit: number analyzed (Participants) | 95
  Glucose, Week 36, < lower limit | 5
  Glucose, Week 52/ withdrawal, > upper limit: number analyzed (Participants) | 114
  Glucose, Week 52/ withdrawal, > upper limit | 45
  Glucose, Week 52/ withdrawal, < lower limit: number analyzed (Participants) | 114
  Glucose, Week 52/ withdrawal, < lower limit | 3
  Creatinine, Baseline, > upper limit | 8
  Creatinine, Baseline, < lower limit | 8
  Creatinine, Week 4, > upper limit: number analyzed (Participants) | 121
  Creatinine, Week 4, > upper limit | 9
  Creatinine, Week 4, < lower limit: number analyzed (Participants) | 121
  Creatinine, Week 4, < lower limit | 8
  Creatinine, Week 12, > upper limit: number analyzed (Participants) | 113
  Creatinine, Week 12, > upper limit | 8
  Creatinine, Week 12, < lower limit: number analyzed (Participants) | 113
  Creatinine, Week 12, < lower limit | 1
  Creatinine, Week 24, > upper limit: number analyzed (Participants) | 106
  Creatinine, Week 24, > upper limit | 9
  Creatinine, Week 24, < lower limit: number analyzed (Participants) | 106
  Creatinine, Week 24, < lower limit | 4
  Creatinine, Week 36, > upper limit: number analyzed (Participants) | 95
  Creatinine, Week 36, > upper limit | 9
  Creatinine, Week 36, < lower limit: number analyzed (Participants) | 95
  Creatinine, Week 36, < lower limit | 3
  Creatinine,Week 52/withdrawal, >upper limit: number analyzed (Participants) | 114
  Creatinine,Week 52/withdrawal, >upper limit | 7
  Creatinine,Week 52/withdrawal, <lower limit: number analyzed (Participants) | 114
  Creatinine,Week 52/withdrawal, <lower limit | 6
  BUN, Baseline, > upper limit | 31
  BUN, Baseline, < lower limit | 1
  BUN, Week 4, > upper limit: number analyzed (Participants) | 121
  BUN, Week 4, > upper limit | 16
  BUN, Week 4, < lower limit: number analyzed (Participants) | 121
  BUN, Week 4, < lower limit | 1
  BUN, Week 12, > upper limit: number analyzed (Participants) | 113
  BUN, Week 12, > upper limit | 23
  BUN, Week 12, < lower limit: number analyzed (Participants) | 113
  BUN, Week 12, < lower limit | 1
  BUN, Week 24, > upper limit: number analyzed (Participants) | 106
  BUN, Week 24, > upper limit | 18
  BUN, Week 36, > upper limit: number analyzed (Participants) | 95
  BUN, Week 36, > upper limit | 21
  BUN, Week 52/ withdrawal, > upper limit: number analyzed (Participants) | 114
  BUN, Week 52/ withdrawal, > upper limit | 22
  BUN, Week 52/ withdrawal, < lower limit: number analyzed (Participants) | 114
  BUN, Week 52/ withdrawal, < lower limit | 1
  UA, Baseline, > upper limit | 35
  UA, Week 4, > upper limit: number analyzed (Participants) | 121
  UA, Week 4, > upper limit | 31
  UA, Week 12, > upper limit: number analyzed (Participants) | 113
  UA, Week 12, > upper limit | 29
  UA, Week 24, > upper limit: number analyzed (Participants) | 106
  UA, Week 24, > upper limit | 19
  UA, Week 36, > upper limit: number analyzed (Participants) | 95
  UA, Week 36, > upper limit | 21
  UA, Week 52/ withdrawal, > upper limit: number analyzed (Participants) | 114
  UA, Week 52/ withdrawal, > upper limit | 32
  Na, Baseline, > upper limit | 2
  Na, Week 4, > upper limit: number analyzed (Participants) | 121
  Na, Week 4, > upper limit | 2
  Na, Week 4, < lower limit: number analyzed (Participants) | 121
  Na, Week 4, < lower limit | 1
  Na, Week 12, > upper limit: number analyzed (Participants) | 113
  Na, Week 12, > upper limit | 2
  Na, Week 24, > upper limit: number analyzed (Participants) | 106
  Na, Week 24, > upper limit | 6
  Na, Week 36, > upper limit: number analyzed (Participants) | 95
  Na, Week 36, > upper limit | 2
  Na, Week 52/ withdrawal, < lower limit: number analyzed (Participants) | 114
  Na, Week 52/ withdrawal, < lower limit | 3
  K, Baseline, > upper limit | 2
  K, Baseline, < lower limit | 1
  K, Week 4, > upper limit: number analyzed (Participants) | 121
  K, Week 4, > upper limit | 2
  K, Week 12, > upper limit: number analyzed (Participants) | 113
  K, Week 12, > upper limit | 4
  K, Week 12, < lower limit: number analyzed (Participants) | 113
  K, Week 12, < lower limit | 2
  K, Week 24, > upper limit: number analyzed (Participants) | 106
  K, Week 24, > upper limit | 3
  K, Week 24, < lower limit: number analyzed (Participants) | 106
  K, Week 24, < lower limit | 2
  K, Week 36, > upper limit: number analyzed (Participants) | 95
  K, Week 36, > upper limit | 7
  K, Week 52/ withdrawal, > upper limit: number analyzed (Participants) | 114
  K, Week 52/ withdrawal, > upper limit | 3
  K, Week 52/ withdrawal, < lower limit: number analyzed (Participants) | 114
  K, Week 52/ withdrawal, < lower limit | 2
  Cl, Baseline, > upper limit | 1
  Cl, Baseline, < lower limit | 1
  Cl, Week 4, > upper limit: number analyzed (Participants) | 121
  Cl, Week 4, > upper limit | 4
  Cl, Week 4, < lower limit: number analyzed (Participants) | 121
  Cl, Week 4, < lower limit | 1
  Cl, Week 12, > upper limit: number analyzed (Participants) | 113
  Cl, Week 12, > upper limit | 2
  Cl, Week 12, < lower limit: number analyzed (Participants) | 113
  Cl, Week 12, < lower limit | 2
  Cl, Week 24, > upper limit: number analyzed (Participants) | 106
  Cl, Week 24, > upper limit | 3
  Cl, Week 24, < lower limit: number analyzed (Participants) | 106
  Cl, Week 24, < lower limit | 2
  Cl, Week 36, > upper limit: number analyzed (Participants) | 95
  Cl, Week 36, > upper limit | 3
  Cl, Week 52/ withdrawal, > upper limit: number analyzed (Participants) | 114
  Cl, Week 52/ withdrawal, > upper limit | 1
  Cl, Week 52/ withdrawal, < lower limit: number analyzed (Participants) | 114
  Cl, Week 52/ withdrawal, < lower limit | 3
  Ca, Baseline, > upper limit | 3
  Ca, Baseline, < lower limit | 2
  Ca, Week 4, > upper limit: number analyzed (Participants) | 121
  Ca, Week 4, > upper limit | 3
  Ca, Week 4, < lower limit: number analyzed (Participants) | 121
  Ca, Week 4, < lower limit | 1
  Ca, Week 12, > upper limit: number analyzed (Participants) | 113
  Ca, Week 12, > upper limit | 3
  Ca, Week 12, < lower limit: number analyzed (Participants) | 113
  Ca, Week 12, < lower limit | 1
  Ca, Week 24, > upper limit: number analyzed (Participants) | 106
  Ca, Week 24, > upper limit | 7
  Ca, Week 36, > upper limit: number analyzed (Participants) | 95
  Ca, Week 36, > upper limit | 4
  Ca, Week 52/ withdrawal, > upper limit: number analyzed (Participants) | 114
  Ca, Week 52/ withdrawal, > upper limit | 3
  Ca, Week 52/ withdrawal, < lower limit: number analyzed (Participants) | 114
  Ca, Week 52/ withdrawal, < lower limit | 1

4. Secondary Outcome: Number of Participants With Abnormal (Shift From Baseline) Urinalysis Parameters
Description: Urinalysis parameters: Urine protein, Glucose and Urobilinogen were presented as shift from Baseline. Only number of participants with urinalysis values more than Baseline values were presented. The plus sign increases with a higher level of glucose and proteins in the urine: 1+: slightly positive, 2+: positive, 3+: high positive and 4+: strongly positive.
Time Frame: Up to Week 56
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GW815SF 50/500 µg
Number analyzed (Participants) | 122
Participants
  Urine protein, Week 4, 1+ to 3+ | 1
  Glucose, Week 4, 3+ to 4+ | 1
  Urine protein, Week 12, 1+ to 2+ | 1
  Urine protein, Week 12, 1+ to 3+ | 1
  Glucose, Week 12, 2+ to 4+ | 1
  Glucose, Week 12, 3+ to 4+ | 1
  Urine protein, Week 24, 1+ to 2+ | 1
  Urine protein, Week 24, 1+ to 3+ | 1
  Glucose, Week 24, 1+ to 2+ | 1
  Glucose, Week 24, 1+ to 4+ | 2
  Glucose, Week 24, 2+ to 4+ | 1
  Urine protein, Week 36, 1+ to 2+ | 1
  Urine protein, Week 36, 1+ to 3+ | 1
  Glucose, Week 36, 1+ to 4+ | 1
  Glucose, Week 36, 2+ to 4+ | 2
  Glucose, Week 36, 3+ to 4+ | 1
  Urine protein, Week 52/withdrawal, 1+ to 3+ | 1
  Glucose, Week 52/withdrawal, 1+ to 2+ | 2
  Glucose, Week 52/withdrawal, 1+ to 4+ | 1
  Glucose, Week 52/withdrawal, 2+ to 4+ | 1

5. Secondary Outcome: Mean Change From Baseline in Level of Plasma Cortisol 1
Description: On each assessment day at Week 24 and 52, adrenal cortical function tests were performed between 8:00-10:00 in the morning. Additional measurements were taken at follow up visit, if the measurements made at Week 52 revealed any abnormalities of clinical significance. Blood samples were taken from participants at rest before undergoing spirometry. Baseline value was the measurement taken at the start of run-in or the treatment period. Change from Baseline was any post Baseline value minus value at Baseline.
Time Frame: Baseline and Week 24 and 52
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micrograms per decilitre (µg/dL)
Arm/Group | GW815SF 50/500 µg
Number analyzed (Participants) | 122
Micrograms per decilitre (µg/dL)
  Week 24: number analyzed (Participants) | 106
  Week 24 | 0.86 (2.945)
  Week 52/Withdrawal: number analyzed (Participants) | 112
  Week 52/Withdrawal | -0.62 (3.118)

6. Secondary Outcome: Mean Level of Plasma Cortisol 2
Description: On each assessment day at Week 24, 52 and follow up, adrenal cortical function tests were performed between 8:00-10:00 in the morning. Additional measurements were taken at follow up visit, if the measurements made at Week 52 revealed any abnormalities of clinical significance. Blood samples were taken from participants at rest before undergoing spirometry.
Time Frame: Up to Week 56
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/dL
Arm/Group | GW815SF 50/500 µg
Number analyzed (Participants) | 122
µg/dL
  Baseline | 9.41 (26.69)
  Week 24: number analyzed (Participants) | 106
  Week 24 | 10.08 (34.19)
  Week 52/Withdrawal: number analyzed (Participants) | 112
  Week 52/Withdrawal | 8.49 (38.63)

7. Secondary Outcome: Mean Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Systolic and diastolic BP was measured in sitting position. Baseline value was the measurement taken at the start of run-in or the treatment period. Change from Baseline was any post Baseline value minus value at Baseline.
Time Frame: Baseline and up to Week 56
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | GW815SF 50/500 µg
Number analyzed (Participants) | 122
Millimeter of mercury (mmHg)
  SBP, Week 4: number analyzed (Participants) | 121
  SBP, Week 4 | 0.5 (14.22)
  SBP, Week 8: number analyzed (Participants) | 118
  SBP, Week 8 | -0.1 (14.74)
  SBP, Week 12: number analyzed (Participants) | 114
  SBP, Week 12 | 0.6 (15.85)
  SBP, Week 16: number analyzed (Participants) | 110
  SBP, Week 16 | 0.7 (15.98)
  SBP, Week 20: number analyzed (Participants) | 107
  SBP, Week 20 | -0.8 (17.08)
  SBP, Week 24: number analyzed (Participants) | 106
  SBP, Week 24 | 0.2 (16.50)
  SBP, Week 28: number analyzed (Participants) | 103
  SBP, Week 28 | -0.4 (17.10)
  SBP, Week 32: number analyzed (Participants) | 97
  SBP, Week 32 | -1.8 (17.74)
  SBP, Week 36: number analyzed (Participants) | 95
  SBP, Week 36 | 1.1 (17.67)
  SBP, Week 40: number analyzed (Participants) | 91
  SBP, Week 40 | 0.4 (17.09)
  SBP, Week 44: number analyzed (Participants) | 89
  SBP, Week 44 | -3.1 (17.48)
  SBP, Week 48: number analyzed (Participants) | 89
  SBP, Week 48 | -4.1 (16.23)
  SBP, Week 52 / withdrawal: number analyzed (Participants) | 119
  SBP, Week 52 / withdrawal | 0.3 (18.12)
  DBP, Week 4: number analyzed (Participants) | 121
  DBP, Week 4 | -0.7 (9.22)
  DBP, Week 8: number analyzed (Participants) | 118
  DBP, Week 8 | -1.2 (9.22)
  DBP, Week 12: number analyzed (Participants) | 114
  DBP, Week 12 | 0.3 (9.72)
  DBP, Week 16: number analyzed (Participants) | 110
  DBP, Week 16 | 0.3 (10.07)
  DBP, Week 20: number analyzed (Participants) | 107
  DBP, Week 20 | -1.4 (9.91)
  DBP, Week 24: number analyzed (Participants) | 106
  DBP, Week 24 | 0.6 (9.88)
  DBP, Week 28: number analyzed (Participants) | 103
  DBP, Week 28 | -0.6 (10.00)
  DBP, Week 32: number analyzed (Participants) | 97
  DBP, Week 32 | -1.4 (11.35)
  DBP, Week 36: number analyzed (Participants) | 95
  DBP, Week 36 | 0.0 (10.16)
  DBP, Week 40: number analyzed (Participants) | 91
  DBP, Week 40 | -1.3 (10.66)
  DBP, Week 44: number analyzed (Participants) | 89
  DBP, Week 44 | -2.1 (11.01)
  DBP, Week 48: number analyzed (Participants) | 89
  DBP, Week 48 | -2.9 (9.44)
  DBP, Week 52 / withdrawal: number analyzed (Participants) | 119
  DBP, Week 52 / withdrawal | -0.1 (10.42)

8. Secondary Outcome: Mean Change From Baseline in Pulse Rate
Description: Pulse rate was measured in sitting position. Baseline value was the measurement taken at the start of run-in or the treatment period. Change from Baseline was any post Baseline value minus value at Baseline.
Time Frame: Baseline and up to Week 56
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: beats per min
Arm/Group | GW815SF 50/500 µg
Number analyzed (Participants) | 122
beats per min
  Week 4: number analyzed (Participants) | 121
  Week 4 | -1.5 (11.19)
  Week 8: number analyzed (Participants) | 118
  Week 8 | -1.6 (10.12)
  Week 12: number analyzed (Participants) | 114
  Week 12 | -0.4 (10.40)
  Week 16: number analyzed (Participants) | 110
  Week 16 | 1.0 (10.03)
  Week 20: number analyzed (Participants) | 106
  Week 20 | 1.1 (11.19)
  Week 24: number analyzed (Participants) | 106
  Week 24 | 1.4 (11.74)
  Week 28: number analyzed (Participants) | 103
  Week 28 | 1.2 (10.23)
  Week 32: number analyzed (Participants) | 97
  Week 32 | 0.4 (10.69)
  Week 36: number analyzed (Participants) | 95
  Week 36 | 0.9 (9.76)
  Week 40: number analyzed (Participants) | 91
  Week 40 | 0.7 (10.94)
  Week 44: number analyzed (Participants) | 89
  Week 44 | 0.4 (11.00)
  Week 48: number analyzed (Participants) | 89
  Week 48 | -0.2 (10.66)
  Week 52 / withdrawal: number analyzed (Participants) | 119
  Week 52 / withdrawal | 0.8 (11.18)

9. Secondary Outcome: Number of Participants With Abnormal Oropharyngeal Examination Findings
Description: Oropharyngeal examination was performed in participants with suspected oral infection (candidiasis).
Time Frame: Up to Week 56
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GW815SF 50/500 µg
Number analyzed (Participants) | 122
Participants
  Week -2 | 1
  Week 0 | 1
  Week 4: number analyzed (Participants) | 121
  Week 4 | 3
  Week 8: number analyzed (Participants) | 118
  Week 8 | 7
  Week 12: number analyzed (Participants) | 114
  Week 12 | 7
  Week 16: number analyzed (Participants) | 110
  Week 16 | 9
  Week 20: number analyzed (Participants) | 107
  Week 20 | 9
  Week 24: number analyzed (Participants) | 106
  Week 24 | 9
  Week 28: number analyzed (Participants) | 103
  Week 28 | 6
  Week 32: number analyzed (Participants) | 97
  Week 32 | 7
  Week 36: number analyzed (Participants) | 95
  Week 36 | 7
  Week 40: number analyzed (Participants) | 91
  Week 40 | 7
  Week 44: number analyzed (Participants) | 89
  Week 44 | 4
  Week 48: number analyzed (Participants) | 89
  Week 48 | 4
  Week52 / withdrawal: number analyzed (Participants) | 119
  Week52 / withdrawal | 8

10. Secondary Outcome: Number of Participants With Abnormal (Clinically Significant) Electrocardiogram (ECG) Findings
Description: On each assessment day at Week 24, 52 and follow up 12-lead ECG was performed. Additional measurements were taken at follow up visit, if the measurements made at Week 52 revealed any abnormalities of clinical significance.
Time Frame: Up to Week 56
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | GW815SF 50/500 µg
Number analyzed (Participants) | 122
Participants
  Baseline | 2
  Week 24 | 3
  Withdrawal | 4

11. Secondary Outcome: Mean Change From Baseline in Bone Mineral Density (BMD)
Description: On each assessment day at Week 52 and follow up, lumber (L1-L4) BMD was determined with a BMD meter by the dual energy X-ray absorption (DEXA) method. Baseline value was the measurement taken during run-in period. Change from Baseline was any value post Baseline minus value at Baseline.
Time Frame: Baseline and up to Week 56
Population: Safety Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per centimeter square
Arm/Group | GW815SF 50/500 µg
Number analyzed (Participants) | 24
Grams per centimeter square | -0.014 (0.0618)

12. Secondary Outcome: Mean Change From Baseline in Weight
Description: Body weight was measured during run-in period, at Week 24 and 52.
Time Frame: Baseline and up to Week 56
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | GW815SF 50/500 µg
Number analyzed (Participants) | 122
Kilograms
  Week 24: number analyzed (Participants) | 106
  Week 24 | 0.17 (1.785)
  Withdrawal: number analyzed (Participants) | 114
  Withdrawal | -0.51 (2.188)

13. Secondary Outcome: Number of Participants With Abnormal (Clinically Significant) Ophthalmological Examinations Findings
Description: On each assessment day at Week 24, 52 and follow up, ophthalmological examinations (vision, cornea, lens, intraocular pressure, fundus oculi) were performed to determine the presence or absence of glaucoma and cataract.
Time Frame: Up to Week 56
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GW815SF 50/500 µg
Number analyzed (Participants) | 122
Participants
  Cataract, Baseline | 3
  Cataract, Week 24 | 2
  Cataract, Withdrawal | 3
  Glaucoma, Baseline | 4
  Glucoma, Week 24 | 4
  Glucoma, Withdrawal | 4

14. Secondary Outcome: Mean Change From Baseline in Peak Expiratory Flow (PEF)
Description: PEF was the maximum speed of expiration measured using spirometer. A participant took rest just before the measurement. At each time of measurement, a participant expired for at least 6 seconds wherever possible. At each time of measurement, at least 3 readings were obtained, and three readings which were obtained in an appropriate manner were stored. Baseline value was the value measured at visit 2. However, when the value at Visit 2 was missing, the value at Visit 1 was used as Baseline. Change from Baseline was any post Baseline value minus Baseline value.
Time Frame: Baseline and up to Week 52
Population: Full analysis set (FAS) Population included all enrolled Population excluding those who had not received investigational product at all and those who had no available data regarding efficacy after starting treatment with investigational product. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Liters per second
Arm/Group | GW815SF 50/500 µg
Number analyzed (Participants) | 122
Liters per second
  Week 4: number analyzed (Participants) | 120
  Week 4 | 0.315 (0.6108)
  Week 8: number analyzed (Participants) | 118
  Week 8 | 0.446 (0.6561)
  Week 12: number analyzed (Participants) | 113
  Week 12 | 0.394 (0.6607)
  Week 16: number analyzed (Participants) | 109
  Week 16 | 0.357 (0.6991)
  Week 20: number analyzed (Participants) | 106
  Week 20 | 0.309 (0.6281)
  Week 24: number analyzed (Participants) | 106
  Week 24 | 0.328 (0.6912)
  Week 28: number analyzed (Participants) | 103
  Week 28 | 0.334 (0.7185)
  Week 32: number analyzed (Participants) | 97
  Week 32 | 0.269 (0.7712)
  Week 36: number analyzed (Participants) | 95
  Week 36 | 0.350 (0.7354)
  Week 40: number analyzed (Participants) | 91
  Week 40 | 0.277 (0.7510)
  Week 44: number analyzed (Participants) | 89
  Week 44 | 0.307 (0.7610)
  Week 48: number analyzed (Participants) | 89
  Week 48 | 0.314 (0.7600)
  Week 52: number analyzed (Participants) | 88
  Week 52 | 0.296 (0.7666)
  Week 52/ withdrawal: number analyzed (Participants) | 106
  Week 52/ withdrawal | 0.229 (0.7942)

15. Secondary Outcome: Mean Change From Baseline in Forced Vital Capacity (FVC)
Description: FVC was the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible measured using spirometer. A participant took rest just before the measurement. At each time of measurement, a participant expired for at least 6 seconds wherever possible. At each time of measurement, at least 3 readings were obtained, and three readings which were obtained in an appropriate manner were stored. Baseline value was the value measured at visit 2. However, when the value at Visit 2 was missing, the value at Visit 1 was used as Baseline. Change from Baseline was any post Baseline value minus Baseline value.
Time Frame: Baseline and up to Week 52
Population: FAS Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | GW815SF 50/500 µg
Number analyzed (Participants) | 122
Liters
  Week 4: number analyzed (Participants) | 120
  Week 4 | 0.128 (0.3048)
  Week 8: number analyzed (Participants) | 118
  Week 8 | 0.156 (0.3411)
  Week 12: number analyzed (Participants) | 113
  Week 12 | 0.142 (0.3772)
  Week 16: number analyzed (Participants) | 109
  Week 16 | 0.140 (0.3199)
  Week 20: number analyzed (Participants) | 106
  Week 20 | 0.106 (0.3318)
  Week 24: number analyzed (Participants) | 106
  Week 24 | 0.127 (0.3247)
  Week 28: number analyzed (Participants) | 103
  Week 28 | 0.149 (0.4115)
  Week 32: number analyzed (Participants) | 97
  Week 32 | 0.142 (0.3587)
  Week 36: number analyzed (Participants) | 95
  Week 36 | 0.147 (0.3447)
  Week 40: number analyzed (Participants) | 91
  Week 40 | 0.148 (0.3803)
  Week 44: number analyzed (Participants) | 89
  Week 44 | 0.156 (0.3699)
  Week 48: number analyzed (Participants) | 89
  Week 48 | 0.147 (0.3713)
  Week 52: number analyzed (Participants) | 88
  Week 52 | 0.170 (0.3841)
  Week 52/ withdrawal: number analyzed (Participants) | 106
  Week 52/ withdrawal | 0.096 (0.4400)

16. Secondary Outcome: Mean Change From Baseline in Maximal Expiratory Flow Rate at 25% (V25) and 50% (V50) of Vital Capacity
Description: V25 and V 50 were measured using spirometer. A participant took rest just before the measurement. At each time of measurement, a participant expired for at least 6 seconds wherever possible. At each time of measurement, at least 3 readings were obtained, and three readings which were obtained in an appropriate manner were stored. Baseline value was the value measured at visit 2. However, when the value at Visit 2 was missing, the value at Visit 1 was used as baseline. Change from Baseline was any post Baseline value minus Baseline value.
Time Frame: Baseline and up to Week 52
Population: FAS Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Liter per second
Arm/Group | GW815SF 50/500 µg
Number analyzed (Participants) | 122
Liter per second
  V25, Baseline: number analyzed (Participants) | 120
  V25, Baseline | 0.018 (0.0595)
  V25, Week 8: number analyzed (Participants) | 118
  V25, Week 8 | 0.021 (0.0685)
  V25, Week 12: number analyzed (Participants) | 113
  V25, Week 12 | 0.015 (0.0611)
  V25, Week 16: number analyzed (Participants) | 109
  V25, Week 16 | 0.016 (0.0713)
  V25, Week 20: number analyzed (Participants) | 106
  V25, Week 20 | 0.012 (0.0693)
  V25, Week 24: number analyzed (Participants) | 106
  V25, Week 24 | 0.017 (0.0649)
  V25, Week 28: number analyzed (Participants) | 103
  V25, Week 28 | 0.012 (0.0753)
  V25, Week 32: number analyzed (Participants) | 97
  V25, Week 32 | 0.009 (0.0628)
  V25, Week 36: number analyzed (Participants) | 95
  V25, Week 36 | 0.018 (0.0689)
  V25, Week 40: number analyzed (Participants) | 91
  V25, Week 40 | 0.022 (0.0715)
  V25, Week 44: number analyzed (Participants) | 89
  V25, Week 44 | 0.015 (0.0681)
  V25, Week 48: number analyzed (Participants) | 89
  V25, Week 48 | 0.010 (0.0735)
  V25, Week 52: number analyzed (Participants) | 88
  V25, Week 52 | 0.017 (0.0839)
  V25, Week 52/ withdrawal: number analyzed (Participants) | 106
  V25, Week 52/ withdrawal | 0.012 (0.0819)
  V50, Week 4: number analyzed (Participants) | 120
  V50, Week 4 | 0.044 (0.1708)
  V50, Week 8: number analyzed (Participants) | 118
  V50, Week 8 | 0.076 (0.1665)
  V50, Week 12: number analyzed (Participants) | 113
  V50, Week 12 | 0.054 (0.1797)
  V50, Week 16: number analyzed (Participants) | 109
  V50, Week 16 | 0.060 (0.1555)
  V50, Week 20: number analyzed (Participants) | 106
  V50, Week 20 | 0.040 (0.1839)
  V50, Week 24: number analyzed (Participants) | 106
  V50, Week 24 | 0.047 (0.1891)
  V50, Week 28: number analyzed (Participants) | 103
  V50, Week 28 | 0.049 (0.1799)
  V50, Week 32: number analyzed (Participants) | 97
  V50, Week 32 | 0.053 (0.1866)
  V50, Week 36: number analyzed (Participants) | 95
  V50, Week 36 | 0.046 (0.1980)
  V50, Week 40: number analyzed (Participants) | 91
  V50, Week 40 | 0.053 (0.1953)
  V50, Week 44: number analyzed (Participants) | 89
  V50, Week 44 | 0.046 (0.1879)
  V50, Week 48: number analyzed (Participants) | 89
  V50, Week 48 | 0.038 (0.1807)
  V50, Week 52: number analyzed (Participants) | 88
  V50, Week 52 | 0.059 (0.2050)
  V50, Week 52/ withdrawal: number analyzed (Participants) | 106
  V50, Week 52/ withdrawal | 0.045 (0.2024)

17. Secondary Outcome: Mean Change From Baseline in Percent of Days Without Use of Rescue Medication
Description: Rescue medication (salbutamol sulfate aerosol provided as an investigational product) was issued to a participant and, when necessary, a spacer at the start of the run-in period. At each time of entry in the Chronic Obstructive Pulmonary Disease (COPD) diary, a participant recorded the number of occasions of rescue medication inhaled in the previous 24 hours in the COPD diary. Baseline was mean value of the consecutive 7 days just before Visit 2. Change from Baseline was any post Baseline value minus Baseline value.
Time Frame: Baseline and up to Week 52
Population: FAS Population.
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | GW815SF 50/500 µg
Number analyzed (Participants) | 122
Percentage of days | 15.6 (33.96)

18. Secondary Outcome: Change From Baseline in Symptom Score With Respect to Breathlessness, Cough, Sputum and Nighttime Awakenings
Description: A participant recorded scores on the scale of 0 to 4 for breathlessness and nighttime awakenings, where 0 indicated no symptoms and 4 indicated severe symptoms; on the scale of 0 to 3 for cough and sputum production, where 0 indicated no symptoms and 3 indicated severe symptoms, in the 24 hours prior to each entry in the COPD diary. Baseline was mean value of the consecutive 7 days just before Visit2. Change from Baseline was any post Baseline value minus Baseline value.
Time Frame: Baseline and up to Week 52
Population: FAS Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GW815SF 50/500 µg
Number analyzed (Participants) | 122
Scores on a scale
  Breathlessness, treatment period | -0.2 (0.57)
  Cough, treatment period | 0.0 (0.51)
  Sputum, treatment period | 0.0 (0.50)
  Nighttime awakenings, treatment period | -0.1 (0.53)

19. Secondary Outcome: Mean Frequency of Moderate and Severe Chronic Obstructive Pulmonary Disease (COPD) Exacerbations
Description: An exacerbation was defined as worsening of the participant's symptoms of cough, sputum production and breathlessness requiring a change in medication. When a moderate or severe COPD exacerbation was observed, details (date of onset, outcome, date of resolution/death, severity, medications provided for treatment, whether the COPD exacerbation required hospitalization, whether the COPD exacerbation required participant withdrawal from the study) were recorded.
Time Frame: Up to Week 56
Population: FAS Population.
Measure: Mean (Standard Deviation); unit: Number of exacerbations
Arm/Group | GW815SF 50/500 µg
Number analyzed (Participants) | 122
Number of exacerbations | 0.456 (1.3560)

20. Secondary Outcome: Mean Observed Maximum Plasma Concentration (Cmax) of Fluticasone Propionate (FP)
Description: For analysis of pharmacokinetic (PK) parameters for FP, blood samples were taken just before dosing (within one hour prior to dosing), 30, 45 minutes, 1, 2, 3, 4, 6, 8 and 12 hours after dosing to determine plasma drug concentrations. The investigational product was taken in fasting condition just before each blood sampling. Parameters were calculated by a model-independent method with the plasma concentration-time profile data in individual participants.
Time Frame: Within one hour prior to dosing, 30, 45 minutes, 1, 2, 3, 4, 6, 8 and 12 hours
Population: All participants evaluable for pharmacokinetic parameters were included in PK Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picograms per milliliter (pg/mL)
Arm/Group | GW815SF 50/500 µg
Number analyzed (Participants) | 12
Picograms per milliliter (pg/mL) | 124.63 (38.597)

21. Secondary Outcome: Mean Cmax of Salmeterol
Description: For analysis of PK parameters for salmeterol, blood samples were taken just before dosing (within one hour prior to dosing), 5, 15, 30, 45 minutes, 1, 2, 3 and 4 hours after dosing to determine plasma drug concentrations. The investigational product was taken in fasting condition just before each blood sampling. Parameters were calculated by a model-independent method with the plasma concentration-time profile data in individual participants.
Time Frame: Within one hour prior to dosing, 5, 15, 30, 45 minutes, 1, 2, 3 and 4 hours
Population: All evaluable subjects. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | GW815SF 50/500 µg
Number analyzed (Participants) | 12
pg/mL | 66.04 (24.955)

22. Secondary Outcome: Median Time of Observed Maximum Plasma Concentration (Tmax) of FP
Description: For analysis of PK parameters for FP, blood samples were taken just before dosing (within one hour prior to dosing), 30, 45 minutes, 1, 2, 3, 4, 6, 8 and 12 hours after dosing to determine plasma drug concentrations. The investigational product was taken in fasting condition just before each blood sampling. Parameters were calculated by a model-independent method with the plasma concentration-time profile data in individual participants.
Time Frame: Within one hour prior to dosing, 30, 45 minutes, 1, 2, 3, 4, 6, 8 and 12 hours
Population: All evaluable subjects. Only those participants with data available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | GW815SF 50/500 µg
Number analyzed (Participants) | 12
hours | 0.875 [0.50 to 4.00]

23. Secondary Outcome: Median Tmax of Salmeterol
Description: as for outcome 21
Time Frame: Within one hour prior to dosing, 5, 15, 30, 45 minutes, 1, 2, 3 and 4 hours
Population: All evaluable subjects. Only those participants with data available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: hour
Arm/Group | GW815SF 50/500 µg
Number analyzed (Participants) | 12
hour | 0.250 [0.08 to 2.00]

24. Secondary Outcome: Mean Area Under the Plasma Concentration-time Curve Over a Dosing Interval [AUC(0-tau)] of FP
Description: as for outcome 22
Time Frame: Within one hour prior to dosing, 30, 45 minutes, 1, 2, 3, 4, 6, 8 and 12 hours
Population: All evaluable subjects. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Hours*picogram per milliliter
Arm/Group | GW815SF 50/500 µg
Number analyzed (Participants) | 12
Hours*picogram per milliliter | 903.48 (303.721)

25. Secondary Outcome: Mean Area Under the Plasma Concentration-time Curve From Zero up to the Last Quantifiable Plasma Concentration [AUC (0-t)] of Salmeterol
Description: as for outcome 21
Time Frame: Within one hour prior to dosing, 5, 15, 30, 45 minutes, 1, 2, 3 and 4 hours
Population: All evaluable subjects. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Hours*picogram per milliliter
Arm/Group | GW815SF 50/500 µg
Number analyzed (Participants) | 10
Hours*picogram per milliliter | 158.16 (81.987)

ADVERSE EVENTS:
Time Frame: All on-treatment AEs and SAEs were assessed up to Week 56
Description: On-treatment AEs and SAEs were reported for Safety Population.
Arm/Group | GW815SF 50/500 µg
All-Cause Mortality (participants affected / at risk) | 2/122
Serious Adverse Events (participants affected / at risk) | 27/122
Other Adverse Events (participants affected / at risk) | 105/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GW815SF 50/500 µg (N=122)
Pneumonia (Infections and infestations) | 10
Atypical mycobacterial infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Oesophageal candidiasis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 9
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Colonic polyp (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Reflux oesophagitis (Gastrointestinal disorders) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vertigo positional (Ear and labyrinth disorders) | 1
Malaise (General disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Atherosclerosis obliterans (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GW815SF 50/500 µg (N=122)
Nasopharyngitis (Infections and infestations) | 59
Oral candidiasis (Infections and infestations) | 22
Bronchitis acute (Infections and infestations) | 12
Pneumonia (Infections and infestations) | 11
Bronchitis (Infections and infestations) | 9
Pharyngitis (Infections and infestations) | 8
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 29
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 17
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 16
Back pain (Musculoskeletal and connective tissue disorders) | 8
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8
Constipation (Gastrointestinal disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.